CLINICAL TRIAL: NCT07324304
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of NWRD06 in Patients With Hepatocellular Carcinoma After Curative Resection.
Brief Title: NWRD06 DNA Plasmid for HCC After Curative Resection.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NWRD06-201
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma; DNA Vaccine; GPC3
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4mg of NWRD06/dose (Experimental)
  Interventions: Biological: NWRD06 administered by electroporation

INTERVENTIONS:
Biological: NWRD06 administered by electroporation — DNA plasmid delivered via IM injection + electroporation using TERESA device

SUMMARY:
This is a single-arm, open-label, multi-center Phase 2 clinical study to evaluate the efficacy and safety of Glypican3 (GPC3)-targeted DNA plasmid vaccine (NWRD06) in patients with GPC3-positive primary hepatocellular carcinoma after curative resection.

DETAILED DESCRIPTION:
Eligible subjects will receive three injections of 4 mg NWRD06 at Weeks 0, 4, and 8. All enrolled subjects will be assessed by tumor imaging at Weeks 12, 24, 36, 48, and 72 after the first dose. These assessments will continue until the first occurrence of any of the following: disease recurrence, meeting withdrawal criteria, initiation of new antitumor therapy, or the completion of Week 72.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years (inclusive), regardless of gender.
2. Histologically or cytologically confirmed diagnosis of hepatocellular carcinoma (HCC).
3. GPC3 positive confirmed by immunohistochemistry (IHC).
4. Barcelona clinic liver cancer (BCLC) stage A/B or Chinese Hepatocellular carcinoma Stage (CNLC) Ib-IIIa.
5. Must have undergone curative treatment (surgical resection or local ablation) for HCC within 12 weeks prior to the first NWRD06 administration; The interval between radical resection and the first NWRD06 administration was less than 12 weeks, and the interval between hepatic artery interventional therapy and the first NWRD06 administration was more than 7 days.
6. No residual intrahepatic lesions, no lymph node metastasis, and no extrahepatic metastasis confirmed by imaging within 4 weeks prior to the first dose.
7. For patients who underwent radical resection, the following intraoperative criteria must be met: 1) No invasion of adjacent organs, no portal lymph node or distant metastasis.

2) Surgical margin negative. 8. No Vp4 macrovascular invasion, hepatic vein or inferior vena cava macrovascular invasion of any grade after radical resection; Notes: Patients with Vp1, Vp2, or Vp3 macrovascular invasion confirmed by imaging or pathology are eligible.

9. ECOG Performance Status of 0 or 1 within 1 week prior to the first dose. 10. Child-Pugh score A/B (≤7) within 1 week prior to the first dose. 11. Adequate organ function within 1 week prior to the first dose: 1) Blood routine: Hemoglobin (Hb) ≥90 g/L; Platelet count (PLT) ≥75×109/L; 2) Liver: Total bilirubin (TB) ≤3× upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN; Plasma albumin ≥30g/L; 3) Coagulation: International Normalized Ratio (INR) ≤2.3. 4) Renal: Serum Creatinine (Scr) ≤1.5 × ULN, OR Creatinine Clearance ≥40 mL/min (if Scr >1.5 × ULN).

12. The expected survival time is more than 6 months; 13. Patients with non-viral primary HCC meet the inclusion criteria. For patients with Hepatitis B virus-related primary HCC(HBV-HCC) or Hepatitis C virus-related primary HCC(HCV-HCC), concurrent antiviral therapy is required.

14. Female subjects of childbearing potential must have a negative serum pregnancy test within 1 week prior to the first dose and must agree to use highly effective contraception from the start of the study treatment until the end of the study. Male subjects must be surgically sterile or must agree to use highly effective contraception during the same period.

15. Have fully understood the study and voluntarily signed the ICF, have good communication with the investigator, and are able to complete all treatments, examinations, and visits stipulated in the study protocol.

Exclusion Criteria:

1. Recurrence or metastasis of HCC prior to the first dose.
2. Has not adequately recovered from toxicities and/or complications of the prior curative procedure.
3. Presence of hepatic encephalopathy.
4. Requires regular renal dialysis.
5. Uncontrolled pleural effusion, pericardial effusion, or clinically significant ascites (defined as ascites not easily controlled by diuretic therapy).
6. History of gastrointestinal bleeding within 28 days prior to screening, or active bleeding, or bleeding tendency.
7. Received any systemic anti-tumor therapy for HCC (including chemotherapy, molecular targeted therapy, bio-immunotherapy) within 28 days prior to screening.
8. Participation in another clinical trial within 28 days prior to screening or still within the observational follow-up period of another trial.
9. Continuous systemic corticosteroid therapy (dose equivalent to >10 mg/day prednisone) for more than one week within 28 days prior to screening (excluding hormone replacement therapy and inhaled corticosteroids).
10. History of immunodeficiency or active autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, etc.).
11. History of allogeneic stem cell, tissue, or solid organ transplantation (including bone marrow transplant).
12. Uncontrolled severe infection (> Grade 2 according to NCI-CTCAE v5.0).
13. Known history of human immunodeficiency virus (HIV) infection or syphilis.
14. Severe dysfunction of other major organs or cardiopulmonary diseases.
15. Epilepsy requiring medication (such as steroids or antiepileptic drugs).
16. History or presence of other malignancies, except for: adequately treated carcinoma in situ of the cervix, basal cell carcinoma of the skin, superficial bladder tumors, ductal carcinoma in situ of the breast, or any other malignancy cured for more than 5 years prior to study entry.
17. Known history of severe allergy, allergic diseases, or allergic constitution.
18. Severe psychiatric disorder.
19. History of drug abuse or alcohol addiction.
20. Pregnant or lactating women, or women with a positive pregnancy test.
21. Any other condition that, in the investigator's judgment, makes the subject unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival rate after treatment with NWRD06 in patients with resected hepatocellular carcinoma. | Week 72
  The number of participants who are recurrence-free at Week 72 after treatment with NWRD06.

SECONDARY OUTCOMES:
Recurrence-free survival after treatment with NWRD06 in patients with resected hepatocellular carcinoma. | up to 72 weeks
  Duration of recurrence-free survival in hepatocellular carcinoma patients after curative resection and treatment with NWRD06.
Incidence and severity of local and systemic adverse events (AEs). | up to 72 weeks
  Based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V5.0, adverse events (AEs) and serious adverse events (SAEs) will be monitored.
Incidence and severity of all serious adverse events (SAEs). | up to 72 weeks
  Incidence and severity of all serious adverse events (SAEs) during the study period (e.g., suspected unexpected serious adverse reactions, unexpected adverse device effects).
Incidence of investigational product-related adverse events (AEs) leading to treatment discontinuation. | up to 72 weeks
  Incidence of AEs leading to discontinuation of study treatment that are related to the investigational product.
Incidence of Grade 3 or higher adverse events (AEs) related to the investigational product. | up to 72 weeks
  Incidence of Grade 3 or higher adverse events (AEs) related to the investigational product.
  Systemic AEs graded per NCI-CTCAE v5.0.
Levels of cellular immune responses. | Weeks 8, 12, 24, 48 and 72
  Levels of cellular immune responses measured by interferon-gamma enzyme-linked immunospot (IFN-γ ELISPOT) assay in peripheral blood mononuclear cells (PBMCs) of subjects at baseline and at weeks 8, 12, 24, 48 and 72 after first dose.
Levels of serum anti-GPC3 antibody titers. | Weeks 8, 12, 24, 48 and 72
  Levels of serum anti-GPC3 antibody titers measured in peripheral blood samples collected at baseline and at weeks 8, 24, and 72 after initial vaccination.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No